CLINICAL TRIAL: NCT07037550
Title: Effectiveness of Strength-based Intervention for Elders With Dementia Living in the Community and Residential Units: a Randomized Controlled Trial
Brief Title: Effectiveness of Strength-based Intervention for Elderly With Dementia Living in the Community
Acronym: STRENGTH-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STRENGTH-B
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Mild Cognitive Impairment; Caregiver; Dementia Alzheimer Type
Keywords: dementia; mild cognitive impairment; caregiver; strength-based intervention; dementia alzheimer type
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The Strength-based intervention incorporates 8-week Ambassador-led strength-based intervention including:
  1. a strength-based assessment to the patient-participant and caregiver done by the Social Worker,
  2. Ambassador-assisted preparation of the strength-based biography,
  3. four Ambassador-led workshops, the workshop will be delivered in group of 6-8 participants by at least 2 Ambassadors, and
  4. one Social Worker-led zoom video conference delivered to the caregivers.
Who Masked: Outcomes Assessor
Masking Description: Another Research Assistant with no information of the random group allocation will execute the posttest assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength-based intervention (Experimental): The Strength-based intervention incorporates 8-week Ambassador-led strength-based intervention including:
  a strength-based assessment to the patient-participant and caregiver done by the Social Worker, Ambassador-assisted preparation of the strength-based biography, four Ambassador-led workshops, the workshop will be delivered in group of 6-8 participants by at least 2 Ambassadors, and one Social Worker-led zoom video conference delivered to the caregivers.
  Interventions: Behavioral: Strength-based intervention
- Usual care (No Intervention): No intervention, continue with usual care

INTERVENTIONS:
Behavioral: Strength-based intervention — The Strength-based intervention incorporates 8-week Ambassador-led strength-based intervention including:
  1. a strength-based assessment to the patient-participant and caregiver done by the Social Worker,
  2. Ambassador-assisted preparation of the strength-based biography,
  3. four Ambassador-led workshops, the workshop will be delivered in group of 6-8 participants by at least 2 Ambassadors, and
  4. one Social Worker-led zoom video conference delivered to the caregivers.
  Arms: Strength-based intervention

SUMMARY:
In the realm of dementia care, the imperative to intervene at the earliest stages of cognitive decline is paramount. Recognizing this pivotal moment, the development of innovative and effective interventions becomes imperative in delaying dementia progression.

Rooted in the Roy Adaptation Model and Zimmer's Theory of Psychological Empowerment, the investigator team has developed the empowerment-based dyadic strength-based intervention, which integrates strength-based and empowerment methodologies. Emphasizing a shift from deficits to capabilities, the strength-based approach fosters awareness of collective strengths within care dyads, facilitating coping mechanisms and resilience in the face of cognitive afflictions.

DETAILED DESCRIPTION:
In the realm of dementia care, the imperative to intervene at the earliest stages of cognitive decline is paramount. Recognizing this pivotal moment, the development of innovative and effective interventions becomes imperative in delaying dementia progression.

Rooted in the Roy Adaptation Model and Zimmer's Theory of Psychological Empowerment, the investigator team has developed the empowerment-based dyadic strength-based intervention, which integrates strength-based and empowerment methodologies. Emphasizing a shift from deficits to capabilities, the strength-based approach fosters awareness of collective strengths within care dyads, facilitating coping mechanisms and resilience in the face of cognitive afflictions.

The objective of this study is:

1. To study the effectiveness of ambassador-led strength-based intervention for patient-participants with dementia living in the community and residential units to enhance their quality of life;
2. To compare how the involvement of young-old volunteers in the strength-based intervention enhance service effectiveness

After obtained the consent baseline data collection will be done. The participants will be randomized to receive either the ambassador-led strength-based intervention of usual care group. The post-test data collection will take place upon the completion of the program (9th week) and at 3-month thereafter.

The Strength-based intervention incorporates 8-week Ambassador-led strength-based intervention including:

1. a strength-based assessment to the patient-participant and caregiver done by the Social Worker,
2. Ambassador-assisted preparation of the strength-based biography,
3. four Ambassador-led workshops, the workshop will be delivered in group of 6-8 participants by at least 2 Ambassadors, and
4. one Social Worker-led zoom video conference delivered to the caregivers.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* a confirmed diagnosis of mild dementia as indicated by the cut-off score of Montreal Cognitive Assessment-5-min at 13-18 for dementia and >18-21 for mild cognitive impairment
* self-reported cognitive complaints
* have the ability to engage in the communication with the research assistant
* able to identify a family caregiver
* consent to participate

Exclusion Criteria:

* person who has communication problems with the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
A battery of cognitive assessments (CAB) | baseline (T0)
  evaluate the global cognition sore by the Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog), the digit span-forward and backward test for attention and working memory, the list learning delayed recall test for episodic memory, 5-min Montreal Cognitive Assessment and Trail-Making Test for complex attention, executive function and task switching. The higher score indicates poor cognitive function
A battery of cognitive assessments (CAB) | 9-weeks immediate posttest (T1)
  evaluate the global cognition sore by the Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog), the digit span-forward and backward test for attention and working memory, the list learning delayed recall test for episodic memory, 5-min Montreal Cognitive Assessment and Trail-Making Test for complex attention, executive function and task switching. The higher score indicates poor cognitive function
A battery of cognitive assessments (CAB) | 3 months after the posttest (T2)
  evaluate the global cognition sore by the Alzheimer's Disease Assessment Scale -Cognitive Subscale (ADAS-Cog), the digit span-forward and backward test for attention and working memory, the list learning delayed recall test for episodic memory, 5-min Montreal Cognitive Assessment and Trail-Making Test for complex attention, executive function and task switching. The higher score indicates poor cognitive function
Quality of Life-Alzheimer's Disease (QoL-AD) | baseline (T0)
  evaluate the health-related quality of life (HRQL) covering physical, functional, psychosocial, interpersonal, and environmental status of the patient with dementia, scales 13 to 52, with higher score indicating better HRQL
Quality of Life-Alzheimer's Disease (QoL-AD) | 9-weeks immediate posttest (T1)
  evaluate the health-related quality of life (HRQL) covering physical, functional, psychosocial, interpersonal, and environmental status of the patient with dementia, scales 13 to 52, with higher score indicating better HRQL
Quality of Life-Alzheimer's Disease (QoL-AD) | 3 months after the posttest (T2)
  evaluate the health-related quality of life (HRQL) covering physical, functional, psychosocial, interpersonal, and environmental status of the patient with dementia, scales 13 to 52, with higher score indicating better HRQL
the 10-item Center for Epidemiologic Studies Depression Scale (CES-D) | baseline (T0)
  evaluate the changes in participant's mood status. The response set is a 4-point Likert scale, scale from 0-30, with a higher score indicating a higher level of depression.
the 10-item Center for Epidemiologic Studies Depression Scale (CES-D) | 9-weeks immediate posttest (T1)
  evaluate the changes in participant's mood status. The response set is a 4-point Likert scale, scale from 0-30, with a higher score indicating a higher level of depression.
the 10-item Center for Epidemiologic Studies Depression Scale (CES-D) | 3 months after the posttest (T2)
  evaluate the changes in participant's mood status. The response set is a 4-point Likert scale, scale from 0-30, with a higher score indicating a higher level of depression.
Dyadic Relationship Scale - Patient version (DRS-patient) | baseline (T0)
  evaluate the quality of interpersonal relationships in the caregiving dyad, in the care recipient perspective. It measures aspects such as communication, support, and satisfaction within the dyad, providing insight into the dynamics of caregiving relationships in dementia care settings. It scale from 0-30 with a higher score indicating a better dyadic relationship.
Dyadic Relationship Scale - Patient version (DRS-patient) | 9-weeks immediate posttest (T1)
  evaluate the quality of interpersonal relationships in the caregiving dyad, in the care recipient perspective. It measures aspects such as communication, support, and satisfaction within the dyad, providing insight into the dynamics of caregiving relationships in dementia care settings. It scale from 0-30 with a higher score indicating a better dyadic relationship.
Dyadic Relationship Scale - Patient version (DRS-patient) | 3 months after the posttest (T2)
  evaluate the quality of interpersonal relationships in the caregiving dyad, in the care recipient perspective. It measures aspects such as communication, support, and satisfaction within the dyad, providing insight into the dynamics of caregiving relationships in dementia care settings. It scale from 0-30 with a higher score indicating a better dyadic relationship.
Dyadic Relationship Scale - Caregiver version (DRS-caregiver) | baseline (T0)
  evaluate the quality of interpersonal relationships in the caregiving dyad, in the caregiver perspective. It measures aspects such as communication, support, and satisfaction within the dyad, providing insight into the dynamics of caregiving relationships in dementia care settings. It scale from 0-33 with a higher score indicating a better dyadic relationship.
Dyadic Relationship Scale - Caregiver version (DRS-caregiver) | 9-weeks immediate posttest (T1)
  evaluate the quality of interpersonal relationships in the caregiving dyad, in the caregiver perspective. It measures aspects such as communication, support, and satisfaction within the dyad, providing insight into the dynamics of caregiving relationships in dementia care settings. It scale from 0-33 with a higher score indicating a better dyadic relationship.
Dyadic Relationship Scale - Caregiver version (DRS-caregiver) | 3 months after the posttest (T2)
  evaluate the quality of interpersonal relationships in the caregiving dyad, in the caregiver perspective. It measures aspects such as communication, support, and satisfaction within the dyad, providing insight into the dynamics of caregiving relationships in dementia care settings. It scale from 0-33 with a higher score indicating a better dyadic relationship.
The Revised Scale for Caregiving Self-Efficacy (RSCSE) | baseline (T0)
  evaluate the perceived self-efficacy in caregiving, to measure the caregivers' perceived self-efficacy in handling the symptoms of the persons with mild cognitive impairment and to control their own emotions. It scale from 0-100 with a higher score indicating a higher caregiving self-efficacy.
The Revised Scale for Caregiving Self-Efficacy (RSCSE) | 9-weeks immediate posttest (T1)
  evaluate the perceived self-efficacy in caregiving, to measure the caregivers' perceived self-efficacy in handling the symptoms of the persons with mild cognitive impairment and to control their own emotions. It scale from 0-100 with a higher score indicating a higher caregiving self-efficacy.
The Revised Scale for Caregiving Self-Efficacy (RSCSE) | 3 months after the posttest (T2)
  evaluate the perceived self-efficacy in caregiving, to measure the caregivers' perceived self-efficacy in handling the symptoms of the persons with mild cognitive impairment and to control their own emotions. It scale from 0-100 with a higher score indicating a higher caregiving self-efficacy.
The Neuro-psychiatric Inventory (NPI) | baseline (T0)
  evaluate the neuro-psychiatric symptoms of the patient with dementia reported by the caregiver, scales from 12 to 96 with higher scores indicating higher severity
The Neuro-psychiatric Inventory (NPI) | 9-weeks immediate posttest (T1)
  evaluate the neuro-psychiatric symptoms of the patient with dementia reported by the caregiver, scales from 12 to 96 with higher scores indicating higher severity
The Neuro-psychiatric Inventory (NPI) | 3 months after the posttest (T2)
  evaluate the neuro-psychiatric symptoms of the patient with dementia reported by the caregiver, scales from 12 to 96 with higher scores indicating higher severity
the Patient-Reported Mild Behavioral Impairment Scale | baseline (T0)
  evaluate the behavioral changes associated with cognitive decline for those with mild cognitive impairment, which enables patients to self-report symptoms, aiding in early detection and intervention for mild behavioral impairment, a potential precursor to dementia. It scale from 0-102 with a higher score indicating a higher risk of behavioral changes associated with cognitive decline.
the Patient-Reported Mild Behavioral Impairment Scale | 9-weeks immediate posttest (T1)
  evaluate the behavioral changes associated with cognitive decline for those with mild cognitive impairment, which enables patients to self-report symptoms, aiding in early detection and intervention for mild behavioral impairment, a potential precursor to dementia. It scale from 0-102 with a higher score indicating a higher risk of behavioral changes associated with cognitive decline.
the Patient-Reported Mild Behavioral Impairment Scale | 3 months after the posttest (T2)
  evaluate the behavioral changes associated with cognitive decline for those with mild cognitive impairment, which enables patients to self-report symptoms, aiding in early detection and intervention for mild behavioral impairment, a potential precursor to dementia. It scale from 0-102 with a higher score indicating a higher risk of behavioral changes associated with cognitive decline.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Haskan Avcı, Ö. (2014). Development of the Dyadic Relationship Scale. Eurasian Journal of Educational Research, 56, 89-108 DOI: http://dx.doi.org/10.14689/ejer.2014.56.6
- [Background] Yu DS, Li PW, Zhang F, Cheng ST, Ng TK, Judge KS. The effects of a dyadic strength-based empowerment program on the health outcomes of people with mild cognitive impairment and their family caregivers: a randomized controlled trial. Clin Interv Aging. 2019 Oct 4;14:1705-1717. doi: 10.2147/CIA.S213006. eCollection 2019. PMID 31686796
- [Background] Yeung PY, Wong LLL, Chan CC, Yung CY, Leung LMJ, Tam YY, Tang LN, Li HS, Lau ML. Montreal Cognitive Assessment - Single Cutoff Achieves Screening Purpose. Neuropsychiatr Dis Treat. 2020 Nov 6;16:2681-2687. doi: 10.2147/NDT.S269243. eCollection 2020. PMID 33192067
- [Background] Smith SC, Lamping DL, Banerjee S, Harwood R, Foley B, Smith P, Cook JC, Murray J, Prince M, Levin E, Mann A, Knapp M. Measurement of health-related quality of life for people with dementia: development of a new instrument (DEMQOL) and an evaluation of current methodology. Health Technol Assess. 2005 Mar;9(10):1-93, iii-iv. doi: 10.3310/hta9100. PMID 15774233
- [Background] Ismail Z, Aguera-Ortiz L, Brodaty H, Cieslak A, Cummings J, Fischer CE, Gauthier S, Geda YE, Herrmann N, Kanji J, Lanctot KL, Miller DS, Mortby ME, Onyike CU, Rosenberg PB, Smith EE, Smith GS, Sultzer DL, Lyketsos C; NPS Professional Interest Area of the International Society of to Advance Alzheimer's Research and Treatment (NPS-PIA of ISTAART). The Mild Behavioral Impairment Checklist (MBI-C): A Rating Scale for Neuropsychiatric Symptoms in Pre-Dementia Populations. J Alzheimers Dis. 2017;56(3):929-938. doi: 10.3233/JAD-160979. PMID 28059789
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Chu LW, Chiu KC, Hui SL, Yu GK, Tsui WJ, Lee PW. The reliability and validity of the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) among the elderly Chinese in Hong Kong. Ann Acad Med Singap. 2000 Jul;29(4):474-85. PMID 11056778
- [Background] Boey KW. Cross-validation of a short form of the CES-D in Chinese elderly. Int J Geriatr Psychiatry. 1999 Aug;14(8):608-17. doi: 10.1002/(sici)1099-1166(199908)14:83.0.co;2-z. PMID 10489651
- [Background] Steffen AM, Gallagher-Thompson D, Arenella KM, Au A, Cheng ST, Crespo M, Cristancho-Lacroix V, Lopez J, Losada-Baltar A, Marquez-Gonzalez M, Nogales-Gonzalez C, Romero-Moreno R. Validating the Revised Scale for Caregiving Self-Efficacy: A Cross-National Review. Gerontologist. 2019 Jul 16;59(4):e325-e342. doi: 10.1093/geront/gny004. PMID 29546334